CLINICAL TRIAL: NCT00006171
Title: A Study of the Effects of Potent Anti-HIV Therapy on Parameters Hypothesized to be Related to the Pathogenesis of Kaposi's Sarcoma (KS) in HIV-Infected Individuals
Brief Title: Effects of Potent Antiretroviral Therapy on Kaposi s Sarcoma
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000193; 00-C-0193; NCT00020319 (obsolete NCT alias)
Record Dates: First submitted 2000-08-10; First posted 2000-08-11 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2012-06-29

CONDITIONS: HIV Seropositivity; Kaposi's Sarcoma; HIV Infections
Keywords: HHV-8; Pathophysiology; AIDS; Cancer; Anti-Retroviral; Kaposi's Sarcoma; HIV
MeSH Terms: conditions — HIV Seropositivity; Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome; Neoplasms

SUMMARY:
Background:

Kaposi s sarcoma (KS) is caused by a gammaherpesvirus called Kaposi s sarcoma-associated herpesvirus (KSHV), or human herpesvirus-8 (HHV-8). However, infection with KSHV is not sufficient to cause KS, and HIV infection is an important cofactor. Treatment of HIV with potent antiretroviral therapy can reduce the risk of KS, and can also induce regression in patients with established HIV-KS. One mechanism by which HIV is believed to contribute to KS is through HIV-induced immunodeficiency which leads to a loss of immunologic control of KSHV and/or KS itself. However, other mechanisms may also contribute.

Objectives:

One primary objective is to assess the effects of the initiation of potent anti-HIV therapy on specific factors possibly linked to the control or pathogenesis of KS, namely serum viral IL-6 and plasma VEGF levels, in patients with KS or at risk for KS by virtue of being infected with KSHV/HHV-8. Another is to assess the effects of anti-HIV therapy on KSHV infection. Secondary objectives are to assess the effects of potent antiretroviral therapy on established KS and other factors related to KS or KSHV infection.

Eligibility:

The principal eligibility factors are age 13 or above, HIV infection, and either KS or infection with KSHV. Exclusion factors include KS that requires specific therapy, recent corticosteroid therapy, recent cytokine therapy, or opportunistic infections requiring therapy.

Design:

Patients will be treated with potent antiretroviral therapy. For patients with established KS, the effects of the therapy on the KS will be monitored. In addition, a variety of factors related to KS, HIV infection, therapy, or KSHV infection will be monitored. These include the HIV viral load, KSHV secretion in saliva, the CD4 count, serum VEGF levels, and serum IL-6 levels.

DETAILED DESCRIPTION:
Background:

Kaposi s sarcoma (KS) is caused by a gammaherpesvirus called Kaposi s sarcoma-associated herpesvirus (KSHV), or human herpesvirus-8 (HHV-8). However, infection with KSHV is not sufficient to cause KS, and HIV infection is an important cofactor. Treatment of HIV with potent antiretroviral therapy can reduce the risk of KS, and can also induce regression in patients with established HIV-KS. One mechanism by which HIV is believed to contribute to KS is through HIV-induced immunodeficiency which leads to a loss of immunologic control of KSHV and/or KS itself. However, other mechanisms may also contribute.

Objectives:

One primary objective is to assess the effects of the initiation of potent anti-HIV therapy on specific factors possibly linked to the control or pathogenesis of KS, namely serum viral IL-6 and plasma VEGF levels, in patients with KS or at risk for KS by virtue of being infected with KSHV/HHV-8. Another is to assess the effects of anti-HIV therapy on KSHV infection. Secondary objectives are to assess the effects of potent antiretroviral therapy on established KS and other factors related to KS or KSHV infection.

Eligibility:

The principal eligibility factors are age 13 or above, HIV infection, and either KS or infection with KSHV. Exclusion factors include KS that requires specific therapy, recent corticosteroid therapy, recent cytokine therapy, or opportunistic infections requiring therapy.

Design:

Patients will be treated with potent antiretroviral therapy. For patients with established KS, the effects of the therapy on the KS will be monitored. In addition, a variety of factors related to KS, HIV infection, therapy, or KSHV infection will be monitored. These include the HIV viral load, KSHV secretion in saliva, the CD4 count, serum VEGF levels, and serum IL-6 levels.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than or equal to 13 years

HIV seropositive

Either a diagnosis of Kaposi's sarcoma and/or HHV-8/KSHV seropositive

EXCLUSION CRITERIA:

Requirement for specific anti-KS therapy

Specific anti-KS therapy within 4 weeks of study entry

Corticosteroid therapy within 4 weeks prior to initiating study

Condition that periodically requires immune suppressive therapy (e.g. asthma)

Cytokine therapy within 4 weeks of study entry

HIV-associated opportunistic complications requiring therapy

Inability to provide informed consent

Investigator recommendation that antiretroviral therapy is in best patient interest

Inability to comply with protocol

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2000-08-07; Study Completion 2012-06-29

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Biggar RJ, Rabkin CS. The epidemiology of AIDS--related neoplasms. Hematol Oncol Clin North Am. 1996 Oct;10(5):997-1010. doi: 10.1016/s0889-8588(05)70380-4. PMID 8880192
- [Background] Goedert JJ, Cote TR, Virgo P, Scoppa SM, Kingma DW, Gail MH, Jaffe ES, Biggar RJ. Spectrum of AIDS-associated malignant disorders. Lancet. 1998 Jun 20;351(9119):1833-9. doi: 10.1016/s0140-6736(97)09028-4. PMID 9652666
- [Background] Martin JN, Ganem DE, Osmond DH, Page-Shafer KA, Macrae D, Kedes DH. Sexual transmission and the natural history of human herpesvirus 8 infection. N Engl J Med. 1998 Apr 2;338(14):948-54. doi: 10.1056/NEJM199804023381403. PMID 9521982